CLINICAL TRIAL: NCT04756024
Title: Determination of Reference Interval of Spot Urinary Oxalate to Creatinine Ratio in Children of Pakistani Origin Under Six Years of Age
Brief Title: Reference Interval of Spot Urinary Oxalate to Creatinine Ratio in Children
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Syed bilal hashmi, Resident, Aga Khan University
Other Study IDs: 2018-0232-345
Record Dates: First submitted 2021-02-15; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Hyperoxaluria
Keywords: Spot oxalate to creatinine ratio; Reference intervals
MeSH Terms: conditions — Hyperoxaluria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reference intervals (RI) of oxalate for the Pakistani population are not readily available. The values used by most labs are usually taken from the literature from studies mainly performed on Caucasian or from the manufacturer package insert of oxalate reagent kits [2]. RI of an analyte assist the clinician in differentiating between health and disease [3]. It is established by testing healthy populations and figuring out what appears to be "normal" for them after defining the reference population demographically. Careful determination and verification or validation of RI by the laboratory are essential to ensure proper utility.

DETAILED DESCRIPTION:
A cross-sectional study was conducted at Section of Chemical Pathology, Department of Pathology and Laboratory Medicine, Aga Khan University, Karachi, from June 2018 to October 2019 after approval from Aga Khan University Hospital's ethical review committee.

Inclusion criteria included children less than six years of age, not suffering from any illness during the last two weeks and no hospitalization since the last four weeks. Children on vitamins or history of kidney stones or family history of kidney stones were excluded.

A standardized questionnaire was used, and recommended target sample size was calculated using CLSI Guidelines C28-A3. Non-probability (consecutive sampling) was done. Parents or guardians of each reference individual were invited to participate in the study. An explanation of the study, consent form (written in the local language, in accordance with the guidelines of the local ethics committee), and the procedure for participation were explained to the parents by the primary investigator. Those who consented were provided with a container for urine collection, and the procedure for the collection was explained. A 5ml random morning urine sample was collected and stored at -30 ºC until analysis after adding 6M hydrochloric acid.

Urinary Oxalate was measured on Micro lab 300 using a kit based on the oxalate oxidase principle by Trinity Biotech Plc, Wicklow, Ireland while creatinine was measured by kinetic Jaffe reaction ADVIA 1800 by Siemens Diagnostic, USA. Samples were analyzed in batches with quality control specimen for validating the results. Oxalate to creatinine ratio (Ox: Cr) was calculated. College of American Pathologist, USA accredits clinical Laboratory of Aga Khan University Hospital.

Data were analyzed by EP evaluator and SPSS 23. Subjects were categorized based on ages into five groups. Group I (0-6 months), Group II (6 months-1 years), Group III (1-2 years), Group IV (2-4 years), and Group V (4-6 years). Descriptive data were analyzed for frequencies and median with IQR. P-value <0.05 was taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included children less than six years of age, not suffering from any illness during the last two weeks and no hospitalization since the last four weeks.

Exclusion Criteria:

* Children on vitamins or history of kidney stones or family history of kidney stones were excluded.

Ages: 15 Days to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children less than 6 years of age (both genders)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Determination of Reference Interval of Spot Urinary Oxalate to Creatinine Ratio in Children of Pakistani Origin Under Six Years of Age | 1 year
  To determine the spot urine oxalate to creatinine reference interval in children under six years of age for our population.

CONTACTS AND LOCATIONS:
Overall Officials: Syed bilal hashmi, MBBS, Principal Investigator — AKUH
Locations (1):
- Syed bilal hashmi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cochat P, Rumsby G. Primary hyperoxaluria. N Engl J Med. 2013 Aug 15;369(7):649-58. doi: 10.1056/NEJMra1301564. No abstract available. PMID 23944302
- [Result] Molla A, Khurshid M, Manser WT, Lalani R, Alam A, Mohammad Z. Suggested reference ranges in clinical chemistry for apparently healthy males and females of Pakistan. J Pak Med Assoc. 1993 Jun;43(6):113-5. PMID 8411612